CLINICAL TRIAL: NCT01551875
Title: A Study to Derive Normative Distribution of CIMT and to Determine Its Correlation With Cardiovascular Risk Factors in Asymptomatic Nationwide Indian Population (SCORE India)
Brief Title: A Study to Derive Normative Distribution of CIMT and to Determine Its Correlation With Cardiovascular Risk Factors
Acronym: Score-India
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CIN-XXX-2011/2; Score-India
Record Dates: First submitted 2012-03-07; First posted 2012-03-13 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Carotid Intima- Media Thickness
Keywords: CIMT; cardiovascular disease; correlation with cardiovascular Risk factors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- subjects who are meeting the inclusion criteria

SUMMARY:
This non-interventional, prospective, multi-centric, cross-sectional study is aimed to obtain the distribution of measurements of CIMT in Indian subjects and will involve approx. 30 investigative sites from all over the country. Each investigative site will be expected to enrol 50 subjects and Carotid intima-media thickness (CIMT) values will be taken for each individual as described in the protocol.

All the procedures could be completed in a single day, however due to any reason any study variable is not taken subject may be asked to come back for a second visit within 7 days of the first visit.

DETAILED DESCRIPTION:
A Study to derive normative distribution of CIMT and to determine its cOrrelation with cardiovascular Risk factors in asymptomatic nationwidE Indian population. (SCORE India)

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent
* Female or male aged 30 years and over

Exclusion Criteria:

* Subjects with established cardiovascular event
* Intake of lipid lowering drug in the past 3 month
* Subjects with known hypersensitivity to carotid bulb
* Pregnant or lactating women

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomatic subjects with or without risk factors but not suffering from any established cardiovascular event.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
CIMT values in centimeters (unit) of male and female subjects without established cardiovascular disease. | at visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Paurus M Irani, MD, Study Director — AstraZeneca Pharma India Ltd.; R R Kasliwal, DM, Principal Investigator — Medanta, The Medicity, Gurgaon
Locations (24):
- India (24):
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Gurgaon, Haryana
  - Research Site, Keshwāpur, Hubli
  - Research Site, Nampally, Hyderabad
  - Research Site, Punjab, Jalanhar
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nerul, Navi Mumbai
  - Research Site, Delhi, New Delhi
  - Research Site, Dhanvantri Nagar, Puducherry
  - Research Site, Jipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Poonkunnam, Thrisur
  - Research Site, Pattom, Trivandum
  - Research Site, Ghaziabad, Uttar Pradesh
  - Research Site, Noida, Uttar Pradesh
  - Research Site, Varanasi, Uttar Pradesh
  - Research Site, Kolkata, West Bengal
  - Research Site, Chandigarh
  - Research Site, Indore
  - Research Site, Lucknow
  - Research Site, Pune